CLINICAL TRIAL: NCT05884112
Title: Treating Comorbid Depression of Patients With Narcolepsy by Intermittent Theta Burst Stimulation: A Preliminary Study
Brief Title: Treating Comorbid Depression of Patients With Narcolepsy by Intermittent Theta Burst Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202102036A3
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-04

CONDITIONS: Narcolepsy
Keywords: hypersomnia; narcolepsy; depression; transcranial magnetic stimulation; neurocognitive function; quality of life
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence; Depression | interventions — Transcranial Magnetic Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participant and doctor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narcolepsy (type1 +type 2) with depression (Experimental): Stimulate with Double 70mm Alpha Coil figure of 8 stimulator (8-shaped stimulator) (Magstim Company, UK, high frequency magnetic stimulator with force power booster), each treatment will give subjects 1800 pulses, including 60 TBS Section stimulation, each section has 2 seconds of stimulation (30 pulses) and 8 seconds of interval, a total stimulation time of 10 minutes.
  Interventions: Device: "MAGSTIM" reprtitive Transcranial Magnetic Stimulator (rTMS) System
- Narcolepsy with depression (Sham Comparator): Sham-control
  Interventions: Device: sham control

INTERVENTIONS:
Device: "MAGSTIM" reprtitive Transcranial Magnetic Stimulator (rTMS) System — iTBS is a new treatment method for depression. It uses the principle of magnetoelectricity to intermittently stimulate local brain nerves. In recent years, domestic and foreign studies have confirmed its efficacy and safety for depression. In addition, research has also It shows that iTBS has better therapeutic effect and efficiency than the previous regular rTMS.
  Arms: Narcolepsy (type1 +type 2) with depression
Device: sham control — sham control
  Arms: Narcolepsy with depression

SUMMARY:
Narcolepsy is a chronic brain disorder. The mechanism is the impairment of brain controlling of sleep and wakefulness. The cause of this disease is still unclear, but common symptoms include excessive day time sleepiness, cataplexy, hypnogogic hallucination, sleep paralysis, and sleep disturbance. Because these symptoms are easily confused together in many situations, it is difficult for doctors to make the diagnosis. Therefore, medical treatment for patients is always delayed. According to previous research report, narcoleptic patients are often delay diagnosis for 10 to 15 years after the onset of the disease. Clearly, to make the diagnosis of narcolepsy is very difficult. Another cause for the delay is the method for diagnosing narcolepsy, which mainly rely on sleep examination instruments and the testing of hypocretin concentration in the cerebrospinal fluid. However, these tests are difficult to carry out in many areas, and diagnosing narcolepsy is still difficult in many countries. To the patients and their families, developing a fast and accurate method or tool for diagnosing narcolepsy is of the utmost importance.

DETAILED DESCRIPTION:
The purposes of this study are as follows: (1) To collect comprehensive narcolepsy and non-narcolepsy brain imaging data. The difference between the two groups will be analyzed. To find the difference between the Type 1 and Type 2 narcolepsy by brain imaging characteristics. Use these data to find the special parameter by "machine learning" and build a predictive model; (2)To collect comprehensive narcolepsy and non-narcolepsy HLA typing data. Attempt to understand the HLA profile of narcoleptic patients and their parents in Taiwan. To analyze the difference between the two groups of Type 1 and Type 2 narcolepsy. Use these data of HLA typing characteristics to find the special parameter by "machine learning" and to establish a predictive model; and (3) categorize and group narcolepsy clinical data, sleep examination data, and the aforementioned data based on machine learning concept and build a predictive model as the basis for developing a fast and accurate" narcolepsy diagnostic tool or model" in the future. Research method: This is a case control study. There are 400 subjects (age 9 - 45) will be collected. These subjects will be divided into the three following groups: (1) experimental group (narcolepsy Type 1, 200 subjects); (2) experimental group (narcolepsy Type 2, 100 subjects); and (3) control group (age and gender matched non-narcolepsy subjects, 100). The investigators will collect all the clinical data for each subject, including clinical characteristics, sleep examination data, actigraphy, HLA typing, and brain imaging data. Data analysis method: the narcolepsy clinical data, sleep examination data, and the aforementioned data were categorized and grouped through data analysis based on computer machine learning, neural network, and predictive model effectiveness analysis concepts. Then the investigators will built a predictive model based on the results.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnosis of Type 1 or Type 2 sleep disorder, and comorbid with depression.
2. The age is introduced between 18-60 years old, regardless of gender.
3. Those who agree to participate in the trial and sign the subject's consent form.

Exclusion Criteria:

1. Combined with epilepsy, brain injury or severe organic brain disease or serious heart disease.
2. Combined with serious other mental disorders, such as bipolar disorder, mental retardation or addiction disorders.
3. Not willing to participate in this study or not willing to fill out the consent form.
4. Those who are not suitable to enter the experiment after being evaluated by PI and co PI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | Screening and following up to six months.
  he Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Below 10 points are non-depressed, 10-18 are mild depression, 19-29 are moderate depression, 30-63 are severe depression.
The Beck Anxiety Inventory | Screening and following up to six months.
  a 21-question method developed by Aaron T. Beck. A multiple-choice self-administered scale designed to measure levels of clinical anxiety that can be used to measure anxiety severity. Takes 5 to 10 minutes to complete. Each answer is scored on a scale of 0 (not at all) to 3 (serious). A higher total score indicates more severe anxiety symptoms. Normalized cut-off values are: 0-7: minimal; 8-15: mild; 16-25: Moderate.

SECONDARY OUTCOMES:
Polysomnography -SE | Screening and following up to six months.
  Change in sleep efficiency (SE, %)based on PSG during the study.
Polysomnography -TST | Screening and following up to six months.
  Change in total sleep time (TST, mins) based on PSG during the study.
Polysomnography -WASO | Screening and following up to six months.
  Change in slow wave sleep (SWS, %) based on PSG during the study.
Polysomnography -REM | Screening and following up to six months.
  Change in REM sleep (%) based on PSG during the study.
Polysomnography -SL | Screening and following up to six months.
  Change in sleep latency (SL, mins) based on PSG during the study.
Polysomnography -SWS | Screening and following up to six months.
  Change in slow wave sleep (SWS, %) based on PSG during the study.
Multiple sleep latency test | Screening and following up to six months.
  Change in Change in sleep latency (SL, mins) based on MSLT during the study.
Conners' Continuous Performance Test | Screening and following up to six months.
  The Conners Continuous Performance Test is a computer administered test that is designed to assess problems with attention.Many statistics are computed including omission errors , commission errors, hit reaction time, hit reaction time standard error, detectability, response style, perseverations , hit reaction time by block, standard error by block, reaction time by ISI , and standard error by ISI. These statistics are converted to T-scores and can be interpreted in terms of various aspects of attention including inattention, impulsivity, and vigilance.Higher rates of correct detections indicate better attentional capacity.
Wisconsin Card Sorting Test | Screening and following up to six months.
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological test that is frequently used to measure such higher-level cognitive processes as attention, perseverance,working memory, abstract thinking and set shifting.
Epworth Sleepoiness Scale | Screening and following up to six months.
  Epworth Sleepoiness Scale (ESS) assesses the responder's propensity to doze or fall asleep during 8 common daily activities, such as: sitting and reading; sitting inactive in a public place; sitting and talking to someone; sitting quietly after a lunch without alcohol; or in a car, while stopped for a few minutes in traffic. An ESS score >10 suggests excessive daytime sleepiness (EDS); ESS score ≥16 suggests a high level of EDS.
Short Form-36 | Screening and following up to six months.
  36-Item Short-Form Health Survey (SF-36) includes 11 major questions that evaluate eight components (0-100), with higher scores indicating better outcome.These components include physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional wellbeing, social functioning, pain, and general health.
PET/MRI | Screening and following up to six months.
  To explore the improvement and difference of narcolepsy and depression symptoms in patients with narcolepsy comorbid depression after rTMS treatment, and to explore the pathological and physiological mechanisms.
Actigraphy-WASO | Screening and following up to six months.
  Wake after sleep onset (WASO) based on actigraphy during the study.
Actigraphy-SE | Screening and following up to six months.
  Sleep efficiency (SE, %) based on actigraphy during the study.
Actigraphy-TST | Screening and following up to six months.
  Total sleep time (TST, mins) based on actigraphy during the study.
Pittsburgh Sleep Quality Index | Screening and following up to six months.
  Nine main questions assess eight sleep components. Assessments included subjective sleep quality, time to sleep, sleep duration, sleep efficiency, sleep disturbances, use of sleeping pills, daytime dysfunction, and global Pittsburgh Sleep Quality Index scores, with higher scores indicating poorer sleep quality.
  Each indicator is scored between 0 and 3. The final composite score is made up of seven combined scores, with a total score ranging from 0 to 21, with lower scores representing healthier sleep quality.
Visual Analogue Scale | Screening and following up to six months.
  Assess the changes in each follow-up of daytime sleepiness and cataplexy symptoms, and the higher the score, the more severe the daytime sleepiness or cataplexy.
  no (0-4 mm), mild (5-44 mm), moderate (45-74 mm), and severe (75-100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shu Huang, PhD, Study Director — Principal Investigator
Locations (1):
- Chang-Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arand D, Bonnet M, Hurwitz T, Mitler M, Rosa R, Sangal RB. The clinical use of the MSLT and MWT. Sleep. 2005 Jan;28(1):123-44. doi: 10.1093/sleep/28.1.123. PMID 15700728
- [Background] Barbey AK, Koenigs M, Grafman J. Dorsolateral prefrontal contributions to human working memory. Cortex. 2013 May;49(5):1195-205. doi: 10.1016/j.cortex.2012.05.022. Epub 2012 Jun 16. PMID 22789779
- [Background] Buskova J, Kemlink D, Ibarburu V, Nevsimalova S, Sonka K. Antidepressants substantially affect basic REM sleep characteristics in narcolepsy-cataplexy patients. Neuro Endocrinol Lett. 2015;36(5):430-3. PMID 26707042
- [Background] Blouin AM, Thannickal TC, Worley PF, Baraban JM, Reti IM, Siegel JM. Narp immunostaining of human hypocretin (orexin) neurons: loss in narcolepsy. Neurology. 2005 Oct 25;65(8):1189-92. doi: 10.1212/01.wnl.0000175219.01544.c8. Epub 2005 Aug 31. PMID 16135770
- [Background] Brooks S, Black J. Novel therapies for narcolepsy. Expert Opin Investig Drugs. 2002 Dec;11(12):1821-7. doi: 10.1517/13543784.11.12.1821. PMID 12457441
- [Background] Corbetta M, Shulman GL. Control of goal-directed and stimulus-driven attention in the brain. Nat Rev Neurosci. 2002 Mar;3(3):201-15. doi: 10.1038/nrn755. PMID 11994752
- [Background] Dauvilliers Y, Arnulf I, Mignot E. Narcolepsy with cataplexy. Lancet. 2007 Feb 10;369(9560):499-511. doi: 10.1016/S0140-6736(07)60237-2. PMID 17292770
- [Background] Nardone R, Bergmann J, Lochner P, Caleri F, Kunz A, Staffen W, Tezzon F, Ladurner G, Trinka E, Golaszewski S. Modafinil reverses hypoexcitability of the motor cortex in narcoleptic patients: a TMS study. Sleep Med. 2010 Oct;11(9):870-5. doi: 10.1016/j.sleep.2010.05.007. PMID 20810311
- [Background] Huang YS, Liu FY, Lin CY, Hsiao IT, Guilleminault C. Brain imaging and cognition in young narcoleptic patients. Sleep Med. 2016 Aug;24:137-144. doi: 10.1016/j.sleep.2015.11.023. Epub 2016 Jan 19. PMID 27663355
- [Background] Huang YS, Hsiao IT, Liu FY, Hwang FM, Lin KL, Huang WC, Guilleminault C. Neurocognition, sleep, and PET findings in type 2 vs type 1 narcolepsy. Neurology. 2018 Apr 24;90(17):e1478-e1487. doi: 10.1212/WNL.0000000000005346. Epub 2018 Mar 30. PMID 29602910
- [Background] Nishino S, Ripley B, Overeem S, Lammers GJ, Mignot E. Hypocretin (orexin) deficiency in human narcolepsy. Lancet. 2000 Jan 1;355(9197):39-40. doi: 10.1016/S0140-6736(99)05582-8. PMID 10615891
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Kales A, Cadieux RJ, Soldatos CR, Bixler EO, Schweitzer PK, Prey WT, Vela-Bueno A. Narcolepsy-cataplexy. I. Clinical and electrophysiologic characteristics. Arch Neurol. 1982 Mar;39(3):164-8. doi: 10.1001/archneur.1982.00510150034008. PMID 7065934
- [Background] Kedzior KK, Gierke L, Gellersen HM, Berlim MT. Cognitive functioning and deep transcranial magnetic stimulation (DTMS) in major psychiatric disorders: A systematic review. J Psychiatr Res. 2016 Apr;75:107-15. doi: 10.1016/j.jpsychires.2015.12.019. Epub 2015 Dec 22. PMID 26828370
- [Background] Lee SA, Kim MK. Effect of Low Frequency Repetitive Transcranial Magnetic Stimulation on Depression and Cognition of Patients with Traumatic Brain Injury: A Randomized Controlled Trial. Med Sci Monit. 2018 Dec 4;24:8789-8794. doi: 10.12659/MSM.911385. PMID 30513530
- [Background] Li CT, Cheng CM, Chen MH, Juan CH, Tu PC, Bai YM, Jeng JS, Lin WC, Tsai SJ, Su TP. Antidepressant Efficacy of Prolonged Intermittent Theta Burst Stimulation Monotherapy for Recurrent Depression and Comparison of Methods for Coil Positioning: A Randomized, Double-Blind, Sham-Controlled Study. Biol Psychiatry. 2020 Mar 1;87(5):443-450. doi: 10.1016/j.biopsych.2019.07.031. Epub 2019 Aug 9. PMID 31563272
- [Background] Mignot E, Hayduk R, Black J, Grumet FC, Guilleminault C. HLA DQB1*0602 is associated with cataplexy in 509 narcoleptic patients. Sleep. 1997 Nov;20(11):1012-20. PMID 9456467
- [Background] Lai JB, Han MM, Xu Y, Hu SH. Effective treatment of narcolepsy-like symptoms with high-frequency repetitive transcranial magnetic stimulation: A case report. Medicine (Baltimore). 2017 Nov;96(46):e8645. doi: 10.1097/MD.0000000000008645. PMID 29145290
- [Background] Naumann A, Daum I. Narcolepsy: pathophysiology and neuropsychological changes. Behav Neurol. 2003;14(3-4):89-98. doi: 10.1155/2003/323060. PMID 14757984
- [Background] Ohayon MM. Narcolepsy is complicated by high medical and psychiatric comorbidities: a comparison with the general population. Sleep Med. 2013 Jun;14(6):488-92. doi: 10.1016/j.sleep.2013.03.002. Epub 2013 May 3. PMID 23643648
- [Background] Ohayon MM, Priest RG, Caulet M, Guilleminault C. Hypnagogic and hypnopompic hallucinations: pathological phenomena? Br J Psychiatry. 1996 Oct;169(4):459-67. doi: 10.1192/bjp.169.4.459. PMID 8894197
- [Background] Posner MI, Petersen SE. The attention system of the human brain. Annu Rev Neurosci. 1990;13:25-42. doi: 10.1146/annurev.ne.13.030190.000325. No abstract available. PMID 2183676
- [Background] Sonmez AI, Kucuker MU, Lewis CP, Kolla BP, Doruk Camsari D, Vande Voort JL, Schak KM, Kung S, Croarkin PE. Improvement in hypersomnia with high frequency repetitive transcranial magnetic stimulation in depressed adolescents: Preliminary evidence from an open-label study. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Mar 8;97:109763. doi: 10.1016/j.pnpbp.2019.109763. Epub 2019 Oct 18. PMID 31634515
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Vijayakumari AA, Khan FR, Varma RP, Radhakrishnan A. Can transcranial magnetic stimulation be used to evaluate patients with narcolepsy? Neurol Sci. 2013 Aug;34(8):1411-20. doi: 10.1007/s10072-012-1253-0. Epub 2012 Nov 29. PMID 23192441
- [Background] Wang W, Chair SY, Thompson DR, Twinn SF. A psychometric evaluation of the Chinese version of the Hospital Anxiety and Depression Scale in patients with coronary heart disease. J Clin Nurs. 2009 Jul;18(13):1908-15. doi: 10.1111/j.1365-2702.2008.02736.x. PMID 19638050
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Yang CM, Huang YS, Song YC. Clinical utility of the Chinese version of the Pediatric Daytime Sleepiness Scale in children with obstructive sleep apnea syndrome and narcolepsy. Psychiatry Clin Neurosci. 2010 Apr;64(2):134-40. doi: 10.1111/j.1440-1819.2009.02054.x. Epub 2010 Feb 1. PMID 20132530